CLINICAL TRIAL: NCT06207292
Title: STereotactic Ablative RadioTherapy in NEWly Synchronous and mEtachRonous (Oligo-persistence, Oligo-induced, Oligo-progression) Oncogene and Non Oncogene Addicted OLIGO-metastatic Non-small Cell Lung Cancer Patients
Brief Title: Stereotactic Ablative Radiotherapy in Synchronous and Metachronous Oligo-Metastatic Non Small Cell Lung Cancer
Acronym: STARTNEWERA-OM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radiotherapy Oncology Centre "Santa Maria" Hospital (Other)
Collaborators: Paola Anselmo,MD (Unknown); Michelina Casale,PhD (Unknown); Fabio Trippa,MD (Unknown)
Responsible Party: Principal Investigator, Fabio Arcidiacono, MD, Principal Investigator, Radiotherapy Oncology Centre "Santa Maria" Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SABR-oligoM NSCLC 810
Record Dates: First submitted 2023-12-27; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: NSCLC; NSCLC Stage IV; Oligometastatic Disease; Non Small Cell Lung Cancer; Non Small Cell Lung Cancer Metastatic; EGF-R Positive Non-Small Cell Lung Cancer; NSCLC Stage IV Without EGFR/ALK Mutation; Non-Small Cell Adenocarcinoma; Non-Small Cell Squamous Lung Cancer; Non-Small Cell Lung Cancer With Mutation in Epidermal Growth Factor Receptor; Synchronous Metastases; Metachronous Metastasis
Keywords: oligo-M NSCLC; SAbR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SABR in oligo-M NSCLC (Experimental): Synchronous and Metachronous oligo-M NSCLC patients will be enrolled to stereotactic ablative radiotherapy (SABR) of primary tumour (T) and/or regional node(s) (N) and oligo-metastatic site (M) with the aim of maintaining ongoing therapy or delaying delaying the start of systemic therapy
  Interventions: Radiation: Stereotactic Ablative Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Ablative Radiotherapy — The prescribed dose of stereotactic ablative radiotherapy (SABR) will be chosen based on the target to be treated and its proximity to organs at risk(s):
  Lung-peripheral 33-45 Gy/ 3 fractions
  Lung-central/ultra-central 35-60 Gy/5 fractions
  Mediastinal/supraclavicular node 35-45 Gy/5 fractions
  Liver 45-54 Gy/3 fractions; 50-65 Gy/5 fractions
  Bone non-spine 30-36 Gy/3 fractions; 35-50 Gy/5 fractions
  Bone spine 30-33 Gy/3 fractions (SIB); 35-40 Gy/ 5 fractions (SIB)
  Abdominal-pelvic node 33-39 Gy/ 3 fractions; 35-50 Gy/5 fractions
  Adrenal gland 30-42 Gy/3 fractions; 35-50 Gy/5 fractions
  Other Names: Targeted Therapy; Immunotherapy; Chemotherapy

SUMMARY:
This is a prospective, non-randomized, single arm, single institution phase II trial to evaluate the safety and effectiveness of stereotactic ablative radiotherapy (SABR) in oncogene addicted and non-oncogene addicted synchronous and/or metachronous oligo-metastatic (oligoM) non-small cell lung cancer (NSCLC) patients.

DETAILED DESCRIPTION:
Targeted Therapies and Immunotherapy have fundamentally changed the treatment of metastatic non-small cell lung cancer (NSCLC).

There is an increasing interest in the use of stereotactic ablative radiotherapy (SABR) for oligo-metastatic (oligo-M) NSCLC patients. It is postulated that definitive treatment of the primary as well as regional node/s and oligo-M in these patients may improve their overall survival (OS). Oligo-M is considered an intermediate state between local and poly-metastatic disease and is commonly defined as 1-5 metastatic lesions, in keeping with the recent European Society of Radiotherapy and Oncology (ESTRO) and American Society for Radiation Oncology (ASTRO) consensus.

If discovered within 4-6months of diagnosis, they are termed synchronous oligo-M. Alternatively, should oligo-M develop following definitive treatment of the primary tumour, this is termed metachronous oligo-M.

Multiple clinical trials have demonstrated prolonged survival following SABR treatment to all sites of oligo-M, particularly in NSCLC.

Targeted therapies (TT) and Immunotherapy (IT) have transformed the landscape of NSCLC treatment by improving OS in metastatic setting. However, most SABR trials for oligo-M patients were conducted in the pre-TT and pre-IT era. How SABR and TT or IT should be integrated in the treatment of oligo-M NSCLC therefore remains an active area of investigation.

Oligo-M is considered a clinically distinct from poly-metastatic disease, presenting a unique therapeutic window during which the treatment of all oligo-M may result in long-term disease control and possibly cure in select cases.

SABR offers the advantages of being non-invasive, safe, and well-tolerated, even by frail patients. It ablates multiple targets simultaneously achieving good rates of local control. The objectives of treating oligo-M using SABR include:

1. ablating all sites of visible disease to reduce tumor burden
2. preventing progression to a poly-metastatic disease state
3. relieving morbidity associated with metastases without a decline in quality of life (QoL)
4. delaying the start of systemic therapy

Reasons to support SABR in oligo-M NSCLC:

1. Systemic treatment alone does not eradicate the presence of all oligo-M disease. SABR may improve local control at the sites of oligo-M decreasing the risk of poly-metastatic widespread by reducing the burden of proliferative malignant cells
2. SABR is a histology-agnostic ablative technique which can eradicate systemic therapy-resistant disease. So, SABR optimizes local control at the sites of oligo-M, thereby delaying the need to start a new systemic therapy or eliminating the morbidity and potential mortality associated with local and eventually distant progression of disease.

   * Targeted therapies (TT) or Immunotherapy (IT) (chemotherapy) will be combined with early SABR of all cancer sites in patients with synchronous oligo-M NSCLC: primary tumour (T), regional node/s (N) and oligo-metastases (M). Eradication of all macroscopic cancer sites at the time of primary diagnosis by combined modality treatment is expected to decrease the risk of resistance development with only microscopic disease potentially remaining. This will result in improvement of progression free survival (PFS), QoL, delayed change of therapy and OS without added high-grade (>G3) toxicity. Synchronous oligo-M NSCLC patients will be enrolled to SABR and TT or IT.
   * Targeted therapies or Immunotherapy (chemotherapy) will be combined with SABR of all cancer residual sites in patients with oligo-persistence, oligo-progressive or oligo- induced oligo-M NSCLC: primary tumour (T), regional node/s (N) and oligo-M. Eradication of all macroscopic cancer sites at the time of oligo-persistence or oligo- progression by combined modality treatment is expected to delay the initiation of a new systemic therapy. This will result in improvement of PFS and QoL, delayed change of therapy and OS without added high-grade (>G3) toxicity. Metachronous oligo-M NSCLC patients will be enrolled to SABR including maintenance TT or IT.
   * Patients unfit for systemic therapy with synchronous or metachronous oligo-M NSCLC will be enrolled to receive SABR alone in all sites of disease. Eradication of all macroscopic cancer sites is expected to delay the widespread and/or symptomatic disease. This will result in improvement of OS and QoL without added high-grade (>G3) toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* histologically confirmed NSCLC
* synchronous oligo-M NSCLC as determined by Positron emission tomography- computed tomography (PET/CT) and brain MRI (AJCC 8th edition)
* metachronous oligo-M NSCLC (oligo-persistence, oligo-progressive, oligo-induced) as determined by PET/CT and brain magnetic resonance imaging (MRI) (AJCC 8th edition)
* patients with at least one target to be treated by SABR at the body
* patients with brain metastases synchronous to the body will be enrolled only if amenable to radiosurgery (the number of brain metastases does not enter into the count of the number of oligo-M)
* patients with a previous history of brain metastases will be enrolled only if the previously treated brain metastases are in control

Exclusion Criteria:

* Ability to understand and the willingness to sign an institutional review board (IRB)- approved informed consent document (either directly or via a legally authorized representative)
* Inability to safely treat target lesions
* Pregnant women are excluded from this study because radiation therapy has known potential for teratogenic or abortifacient effects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2024-01 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
new systemic therapy-free survival | 6 months; 1 year, 2 years, 3 years and 5 years
  time that the patient maintains the same therapy without the need to change it
systemic therapy-free survival | 6 months; 1 year, 2 years, 3 years and 5 years
  time in which the patient does not need to start systemic therapy (for patients without active systemic therapy)
proportion of patients experiencing grade 3 or higher toxicities | 6 months; 1 year, 2 years, 3 years and 5 years
  SABR will be considered safe if no grade (G) or higher toxicities appears. Toxicity will be evaluated according CTCAE scale

SECONDARY OUTCOMES:
progression free survival | 6 months; 1 year, 2 years, 3 years and 5 years
  The interval between treatment and radiological evidence of any progression
overall survival | 6 months; 1 year, 2 years, 3 years and 5 years
  The interval between treatment and death
local control | 6 months; 1 year, 2 years, 3 years and 5 years
  A lack of progression (i.e. any response and stable disease) of the treated volume
time to new oligo-metastatic evidence | 6 months; 1 year, 2 years, 3 years and 5 years
  The interval between treatment and radiological evidence of new oligo-metastatic progression amenable by SABR
time to time to poly-metastatic progression not amenable by SABR | 6 months; 1 year, 2 years, 3 years and 5 years
  The interval between treatment and radiological evidence of poly-metastatic progression not amenable by SABR

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Arcidiacono, MD, Principal Investigator — Radiotherapy Oncology Centre "S.Maria" Hospital, Terni; Paola Anselmo, MD, Principal Investigator — Radiotherapy Oncology Centre "S.Maria" Hospital, Terni; Michelina Casale, PhD, Principal Investigator — Radiotherapy Oncology Centre "S.Maria" Hospital, Terni; Fabio Trippa, MD, Study Director — Radiotherapy Oncology Centre "S.Maria" Hospital, Terni
Locations (1):
- Radiotherapy Oncology Centre "S.Maria" Hospital, Terni, TR, Italy

REFERENCES:
- [Result] Guckenberger M, Lievens Y, Bouma AB, Collette L, Dekker A, deSouza NM, Dingemans AC, Fournier B, Hurkmans C, Lecouvet FE, Meattini I, Mendez Romero A, Ricardi U, Russell NS, Schanne DH, Scorsetti M, Tombal B, Verellen D, Verfaillie C, Ost P. Characterisation and classification of oligometastatic disease: a European Society for Radiotherapy and Oncology and European Organisation for Research and Treatment of Cancer consensus recommendation. Lancet Oncol. 2020 Jan;21(1):e18-e28. doi: 10.1016/S1470-2045(19)30718-1. PMID 31908301
- [Result] Lievens Y, Guckenberger M, Gomez D, Hoyer M, Iyengar P, Kindts I, Mendez Romero A, Nevens D, Palma D, Park C, Ricardi U, Scorsetti M, Yu J, Woodward WA. Defining oligometastatic disease from a radiation oncology perspective: An ESTRO-ASTRO consensus document. Radiother Oncol. 2020 Jul;148:157-166. doi: 10.1016/j.radonc.2020.04.003. Epub 2020 Apr 22. PMID 32388150
- [Result] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Griffioen G, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Bauman GS, Warner A, Senan S. Stereotactic ablative radiotherapy versus standard of care palliative treatment in patients with oligometastatic cancers (SABR-COMET): a randomised, phase 2, open-label trial. Lancet. 2019 May 18;393(10185):2051-2058. doi: 10.1016/S0140-6736(18)32487-5. Epub 2019 Apr 11. PMID 30982687
- [Result] Palma DA, Olson R, Harrow S, Gaede S, Louie AV, Haasbeek C, Mulroy L, Lock M, Rodrigues GB, Yaremko BP, Schellenberg D, Ahmad B, Senthi S, Swaminath A, Kopek N, Liu M, Moore K, Currie S, Schlijper R, Bauman GS, Laba J, Qu XM, Warner A, Senan S. Stereotactic Ablative Radiotherapy for the Comprehensive Treatment of Oligometastatic Cancers: Long-Term Results of the SABR-COMET Phase II Randomized Trial. J Clin Oncol. 2020 Sep 1;38(25):2830-2838. doi: 10.1200/JCO.20.00818. Epub 2020 Jun 2. PMID 32484754
- [Result] Correa RJ, Salama JK, Milano MT, Palma DA. Stereotactic Body Radiotherapy for Oligometastasis: Opportunities for Biology to Guide Clinical Management. Cancer J. 2016 Jul-Aug;22(4):247-56. doi: 10.1097/PPO.0000000000000202. PMID 27441744
- [Result] Iyengar P, Wardak Z, Gerber DE, Tumati V, Ahn C, Hughes RS, Dowell JE, Cheedella N, Nedzi L, Westover KD, Pulipparacharuvil S, Choy H, Timmerman RD. Consolidative Radiotherapy for Limited Metastatic Non-Small-Cell Lung Cancer: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2018 Jan 11;4(1):e173501. doi: 10.1001/jamaoncol.2017.3501. Epub 2018 Jan 11. PMID 28973074
- [Result] Gomez DR, Tang C, Zhang J, Blumenschein GR Jr, Hernandez M, Lee JJ, Ye R, Palma DA, Louie AV, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Welsh JW, Gibbons DL, Karam JA, Kavanagh BD, Tsao AS, Sepesi B, Swisher SG, Heymach JV. Local Consolidative Therapy Vs. Maintenance Therapy or Observation for Patients With Oligometastatic Non-Small-Cell Lung Cancer: Long-Term Results of a Multi-Institutional, Phase II, Randomized Study. J Clin Oncol. 2019 Jun 20;37(18):1558-1565. doi: 10.1200/JCO.19.00201. Epub 2019 May 8. PMID 31067138
- [Result] Wang XS, Bai YF, Verma V, Yu RL, Tian W, Ao R, Deng Y, Zhu XQ, Liu H, Pan HX, Yang L, Bai HS, Luo X, Guo Y, Zhou MX, Sun YM, Zhang ZC, Li SM, Cheng X, Tan BX, Han LF, Liu YY, Zhang K, Zeng FX, Jia L, Hao XB, Wang YY, Feng G, Xie K, Lu Y, Zeng M. Randomized Trial of First-Line Tyrosine Kinase Inhibitor With or Without Radiotherapy for Synchronous Oligometastatic EGFR-Mutated Non-Small Cell Lung Cancer. J Natl Cancer Inst. 2023 Jun 8;115(6):742-748. doi: 10.1093/jnci/djac015. PMID 35094066
- [Result] Peng P, Gong J, Zhang Y, Zhou S, Li Y, Han G, Meng R, Chen Y, Yang M, Shen Q, Chu Q, Xia S, Zhang P, Zhang L, Chen Y, Zhang L. EGFR-TKIs plus stereotactic body radiation therapy (SBRT) for stage IV Non-small cell lung cancer (NSCLC): A prospective, multicenter, randomized, controlled phase II study. Radiother Oncol. 2023 Jul;184:109681. doi: 10.1016/j.radonc.2023.109681. Epub 2023 Apr 25. PMID 37105304
- [Result] Arcidiacono F, Anselmo P, Casale M, Zannori C, Ragusa M, Mancioli F, Marchetti G, Loreti F, Italiani M, Bracarda S, Maranzano E, Trippa F. STereotactic Ablative RadioTherapy in NEWly Diagnosed and Recurrent Locally Advanced Non-Small Cell Lung Cancer Patients Unfit for ConcurrEnt RAdio-Chemotherapy: Early Analysis of the START-NEW-ERA Non-Randomised Phase II Trial. Int J Radiat Oncol Biol Phys. 2023 Mar 15;115(4):886-896. doi: 10.1016/j.ijrobp.2022.10.025. Epub 2022 Oct 24. PMID 36288758
- [Result] Bahig H, Tonneau M, Blais N, Wong P, Filion E, Campeau MP, Vu T, Al-Saleh A, Tehfe M, Florescu M, Roberge D, Masucci L, Richard C, Menard C, Routy B. Stereotactic Ablative Radiotherapy for oligo-progressive disease refractory to systemic therapy in Non-Small Cell Lung Cancer: A registry-based phase II randomized trial (SUPPRESS-NSCLC). Clin Transl Radiat Oncol. 2022 Jan 5;33:115-119. doi: 10.1016/j.ctro.2021.12.008. eCollection 2022 Mar. PMID 35243022
- [Result] Jongbloed M, Bartolomeo V, Steens M, Dursun S, van de Lisdonk T, De Ruysscher DKM, Hendriks LEL. Treatment outcome of patients with synchronous oligometastatic non-small cell lung cancer in the immunotherapy era: Analysis of a real-life intention-to-treat population. Eur J Cancer. 2023 Sep;190:112947. doi: 10.1016/j.ejca.2023.112947. Epub 2023 Jun 20. PMID 37451182
- [Result] Remon J, Menis J, Levy A, De Ruysscher DKM, Hendriks LEL. How to optimize the incorporation of immunotherapy in trials for oligometastatic non-small cell lung cancer: a narrative review. Transl Lung Cancer Res. 2021 Jul;10(7):3486-3502. doi: 10.21037/tlcr-20-1065. PMID 34430382
- [Result] Zayed S, Louie AV, Breadner DA, Palma DA, Correa RJM. Radiation and immune checkpoint inhibitors in the treatment of oligometastatic non-small-cell lung cancer: a practical review of rationale, recent data, and research questions. Ther Adv Med Oncol. 2023 Jul 8;15:17588359231183668. doi: 10.1177/17588359231183668. eCollection 2023. PMID 37435562
- [Result] Baydoun A, Lee VL, Biswas T. Oligometastatic Non-Small Cell Lung Cancer: A Practical Review of Prospective Trials. Cancers (Basel). 2022 Oct 29;14(21):5339. doi: 10.3390/cancers14215339. PMID 36358757
- [Result] Wahl RL, Jacene H, Kasamon Y, Lodge MA. From RECIST to PERCIST: Evolving Considerations for PET response criteria in solid tumors. J Nucl Med. 2009 May;50 Suppl 1(Suppl 1):122S-50S. doi: 10.2967/jnumed.108.057307. PMID 19403881
- [Result] Arcidiacono F, Aristei C, Marchionni A, Italiani M, Fulcheri CPL, Saldi S, Casale M, Ingrosso G, Anselmo P, Maranzano E. Stereotactic body radiotherapy for adrenal oligometastasis in lung cancer patients. Br J Radiol. 2020 Nov 1;93(1115):20200645. doi: 10.1259/bjr.20200645. Epub 2020 Sep 2. PMID 32822540